CLINICAL TRIAL: NCT03122457
Title: Improvement of Perimenstrual Acne With Clindamycin Phosphate and Benzoyl Peroxide 1.2%/3.75% Combination Gel
Brief Title: Perimenstrual Acne With Clindamycin Phosphate and Benzoyl Peroxide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Anjali Vekaria, Chief Resident, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-1230
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Benzoyl Peroxide

STUDY DESIGN:
Intervention Model Description: Application of clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel to treat perimenstrual acne
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lidamycin phosphate and benzoyl peroxide 1.2%/3.75% combo (Experimental): lidamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel; daily use for 99 days
  Interventions: Drug: lidamycin phosphate and benzoyl peroxide 1.2%/3.75% combination

INTERVENTIONS:
Drug: lidamycin phosphate and benzoyl peroxide 1.2%/3.75% combination — At Day 15, patients will be re-assessed and dispensed the investigational product and instructed on its daily use. Patients will continue to return every 14 days to have their skin assessed until their final visit on day 99, one week after their 3rd menses on treatment (4th menses on study).

SUMMARY:
The study team plans to enroll a total of 40 subjects with self-reported perimenstrual acne. Eligible women will be over the age of 18 and not on any current therapy. The patients will first arrive for a screening visit, where they will be given questionnaires on acne quality of life (acne QOL) and subjective assessments as well as flare ups (as used in the study by Geller et al). The patients' skin will be assessed for inflammatory and non-inflammatory acne vulgaris. The baseline visit (day 1) will be scheduled for one week prior to the first day of menses (as studies indicate that most women have their acne flare during this time). The study team will perform a zit count (counting papules, pustules, and comedones) and global assessment, and the patient will be instructed to record their menses (which they will do for the duration of the study). The patients will then return in 2 weeks, at day 15, and they will be re-assessed. The patients will be dispensed the investigational product and instructed on its daily use. The patients will continue to return every 14 days to have their skin assessed until their final visit on day 99, one week after their 3rd menses on treatment (4th menses on study). The duration of the study per patient is approximately 4 months, and the study team anticipates an enrollment period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* Women who have had their first menses at least 12 months ago, and who currently have regular menses.
* Subjects must be able to read and understand English, and be able and willing to complete the survey.
* Subjects must have a self-reported complaint of peri-menstrual acne which has occurred monthly for the last 6 months.
* Subjects must be willing to forego any other therapy to the treatment area for the duration of the study.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* Subjects must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.
* Subjects must be willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant, Depo-Provera, double barrier methods (e.g., condom and spermicide) and abstinence.

Exclusion Criteria:

* Male subjects.
* Post-menopausal women.
* Women who do not suffer from acne.
* Subjects who are allergic to clindamycin, benzoyl peroxide, lidocaine or any other ingredients listed in the study medication.
* Subjects with an unstable medical condition as deemed by the clinical investigator.
* Subjects with ulcerative colitis or Crohn's disease.
* Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of acne.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have used any topical prescription medications on the study area within 30 days prior to Visit 2 / Baseline.
* Subjects on a stable dose of oral contraceptives for less than 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Shroff, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from July 2015 through August 2019 Please confirm the date of the first enrollment (month, day, year) Please confirm the date of the last study visit or the last date that data was collected (month, day, year)
Period: Overall Study
Arm/Group | Lidamycin Phosphate and Benzoyl Peroxide 1.2%/3.75% Combo
Started | 22
Completed | 16
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lidamycin Phosphate and Benzoyl Peroxide 1.2%/3.75% Combo
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: PGA Score
Description: Treatment Success defined as a score of 0 (clear) to 1 (almost clear) at day 99 (final study visit) by acne PGA scoring system. Full PGA scale from 0-5, with lower score indicating better drug efficacy
Time Frame: Day 99
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lidamycin Phosphate and Benzoyl Peroxide 1.2%/3.75% Combo
Number analyzed (Participants) | 22
score on a scale | 0.53 (0.29)

2. Secondary Outcome: Adverse Event Severity
Description: Safety/drug-tolerance evaluated by subject-reported adverse events as well as physician evaluated erythema, scaling, drying, and stinging/burning on a 0-3 point scale, where 0=none and 3=severe.
Time Frame: Day 99
Measure: Count of Participants; unit: Participants
Arm/Group | Lidamycin Phosphate and Benzoyl Peroxide 1.2%/3.75% Combo
Number analyzed (Participants) | 22
Participants
  0 | 22
  1 | 0
  2 | 0
  3 | 0

ADVERSE EVENTS:
Time Frame: 99 days
Arm/Group | Lidamycin Phosphate and Benzoyl Peroxide 1.2%/3.75% Combo
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03122457/Prot_SAP_000.pdf